CLINICAL TRIAL: NCT00717730
Title: Routine Administration of Folic Acid and Vitamin B12 to Prevent Childhood Infections in Young Indian Children
Brief Title: Folic Acid and Vitamin B12 in Young Indian Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tor A. Strand (Other)
Collaborators: Society for Essential Health Action and Training, New Delhi, India (Unknown); Thrasher Research Fund (Other)
Responsible Party: Sponsor-Investigator, Tor A. Strand, Professor II, Centre For International Health
Organization: Centre For International Health (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RCN172226
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Diarrhea; Pneumonia
Keywords: Nutrition; Children; Folate; Vitamin B12; India; Homocysteine; Methyl Malonic Acid
MeSH Terms: conditions — Diarrhea; Pneumonia | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Placebo Comparator): Placebo dietary supplement
  Interventions: Dietary Supplement: Placebo
- B (Experimental): Folic acid
  Interventions: Dietary Supplement: Folic Acid
- C (Experimental): Vitamin B12
  Interventions: Dietary Supplement: Vitamin B12
- D (Experimental): Folic acid and Vitamin B12
  Interventions: Dietary Supplement: Folic acid and vitamin B12

INTERVENTIONS:
Dietary Supplement: Folic Acid — 150µgm/day for 6 months in children older than 11 months and 80µgm in 6 to 11 months.
  Other Names: Folate
  Arms: B
Dietary Supplement: Vitamin B12 — 1.8µgm/day for 6 months in children older than 11 months and 0.5µgm in 6 to 11 months.
  Other Names: Cobalamin
  Arms: C
Dietary Supplement: Placebo — Placebo with no active ingredients
  Arms: A
Dietary Supplement: Folic acid and vitamin B12 — Folic acid 150µgm/day for 6 months in children older than 11 months and 80µgm in 6 to 11 months vitamin B12 1.8µgm/day for 6 months in children older than 11 months and 0.5µgm in 6 to 11 months.
  Arms: D

SUMMARY:
Hypothesis: Supplementation of two recommended daily allowances (RDA) of folic acid with or without simultaneous administration of vitamin B12 reduces the rates of acute lower respiratory tract infections (ALRI), clinical pneumonia and diarrhea.

Design/Methods We will conduct a preventive randomized placebo controlled clinical trial of folic acid and vitamin B12 supplementation in 1000 children aged 6 to 30 months living in a low to middle-income socioeconomic setting in New Delhi, India. Children aged 6-30 months will be identified through a survey. Eligible and willing Children aged 6-30 months will be randomized to 4 treatment groups. Trial to enrollment informed consent will be obtained by the Study Physician/Supervisor. At enrollment a baseline form will be filled and the child weight and length taken. The baseline blood samples will be collected. The supplements will be given daily for 6 months. Morbidity will be ascertained through biweekly home visits by field workers.

DETAILED DESCRIPTION:
Pneumonia and diarrhea are among the leading causes of poor health and death in young children of developing countries.

Many of these children have inadequate intakes of several vitamins and minerals. Folate and vitamin B12 are important for normal function of the immune system. Deficiencies of these vitamins are often part of general malnutrition and might be responsible for the excess morbidity and mortality seen in malnourished children. In a recent cohort study in almost 2,500 Indian children we demonstrated that those with poor folate status had higher rates of diarrhea and pneumonia. This study also showed that children that were not breastfed had poor folate status and our analyses suggested that the effect of breastfeeding in preventing respiratory and gastrointestinal infections could be explained by the folate content of breast milk. The finding that poor folate status is related to increased susceptibility to childhood infections needs to be confirmed in well conducted clinical trials in populations where folate deficiency is prevalent.

This trial aims to examine whether daily supplementation of 2 recommended doses of folate or vitamin B12 or both will lessen the incidence of acute lower respiratory tract infections and diarrhea. We will also measure if the supplementation improves the weight and length of supplemented children.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 to 30 months
* Either sex
* Likely to reside in area for next 6 months

Exclusion Criteria:

* Severe systemic illness requiring hospitalization
* Severe malnutrition, i.e. weight for height < -3 z of the WHO standard for this age group. For ethical reasons these children require micronutrient supplementation and adequate medical care.
* Non consent
* Consuming vitamin supplements that include folic acid and vitamin B12.
* Severe anemia (Hb < 7 g/dL).

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of episodes diarrhea (all, severe, prolonged) and pneumonia (ALRI, Clinical pneumonia) | 6 months
Prevalence of diarrhea | 6 months

SECONDARY OUTCOMES:
Growth (length for age, weight for age, and length for weight) | 6 month
Adverse events (vomiting and gastric discomfort) | 6 months
Changes in folate, vitamin B12, methyl malonic acid, and homocysteine concentration | 6 months
Developmental Milestones | End study, i.e. after 6 months of vitamin B12 and/or folic acid administration
  Developmental milestones. The developmental milestones will be measured using the ASQ-3. ASQ-3 is an easily administered and comprehensive checklist consisting of 30 items measuring skills in 5 different domains; Communication, Gross Motor, Fine Motor, Personal-Social and Problem-Solving. The questionnaires are divided into two-month intervals for use with children 4-60 months of age, and scores are normed to indicate whether children are developing age-appropriately.
Measure the association between pneumonia incidence and the plasma mannose binding lectin (MBL) concentration | Baseline blood samples
Measure the exposure to Cryptosporidium spp | Baseline blood samples
  We will measure the exposure to Cryptosporidium spp. in Indian children aged 6-30 months by measurement of antibodies to recombinant gp15, a conserved surface protein in plasma samples taken at baseline.
Measure the association between the antibody response to Cryptosporidium and plasma MBL | Baseline blood samples
Compare the change in plasma MBL between the intervention groups | 6 months
  We will compare the change in plasma MBL between those who have been given 2 RDA of vitamin B12 and/or folic acid with those who were given placebo in a subsample of 256 children.
Vitamin D status | Baseline blood samples
  We will measure vitamin D (25-hydroxy vitamin D) in all children at baseline to describe the vitamin D status and the proportion with vitamin D deficiency.
Vitamin D status and the risk for respiratory infections | Baseline samples and 6 months follow up
  We will measure the vitamin D status at baseline and assess to what extent it predicts the risk of subsequent respiratory tract infections over the next 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, MD, PhD, Principal Investigator — University of Bergen; Sunita Taneja, MBBS, PhD, Principal Investigator — Society for Essential Health Action and Training
Locations (1):
- Society for Essential Health Action and Training, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Taneja S, Bhandari N, Strand TA, Sommerfelt H, Refsum H, Ueland PM, Schneede J, Bahl R, Bhan MK. Cobalamin and folate status in infants and young children in a low-to-middle income community in India. Am J Clin Nutr. 2007 Nov;86(5):1302-9. doi: 10.1093/ajcn/86.5.1302. PMID 17991639
- [Background] Strand TA, Taneja S, Bhandari N, Refsum H, Ueland PM, Gjessing HK, Bahl R, Schneede J, Bhan MK, Sommerfelt H. Folate, but not vitamin B-12 status, predicts respiratory morbidity in north Indian children. Am J Clin Nutr. 2007 Jul;86(1):139-44. doi: 10.1093/ajcn/86.1.139. PMID 17616773
- [Background] Allen LH. Multiple micronutrients in pregnancy and lactation: an overview. Am J Clin Nutr. 2005 May;81(5):1206S-1212S. doi: 10.1093/ajcn/81.5.1206. PMID 15883453
- [Background] Smith AD, Kim YI, Refsum H. Is folic acid good for everyone? Am J Clin Nutr. 2008 Mar;87(3):517-33. doi: 10.1093/ajcn/87.3.517. PMID 18326588
- [Background] Sazawal S, Dhingra U, Dhingra P, Hiremath G, Kumar J, Sarkar A, Menon VP, Black RE. Effects of fortified milk on morbidity in young children in north India: community based, randomised, double masked placebo controlled trial. BMJ. 2007 Jan 20;334(7585):140. doi: 10.1136/bmj.39035.482396.55. Epub 2006 Nov 28. PMID 17132678
- [Background] Tielsch JM, Khatry SK, Stoltzfus RJ, Katz J, LeClerq SC, Adhikari R, Mullany LC, Shresta S, Black RE. Effect of routine prophylactic supplementation with iron and folic acid on preschool child mortality in southern Nepal: community-based, cluster-randomised, placebo-controlled trial. Lancet. 2006 Jan 14;367(9505):144-52. doi: 10.1016/S0140-6736(06)67963-4. PMID 16413878
- [Background] Fawzi WW, Msamanga GI, Spiegelman D, Urassa EJ, McGrath N, Mwakagile D, Antelman G, Mbise R, Herrera G, Kapiga S, Willett W, Hunter DJ. Randomised trial of effects of vitamin supplements on pregnancy outcomes and T cell counts in HIV-1-infected women in Tanzania. Lancet. 1998 May 16;351(9114):1477-82. doi: 10.1016/s0140-6736(98)04197-x. PMID 9605804
- [Background] Sazawal S, Black RE, Ramsan M, Chwaya HM, Stoltzfus RJ, Dutta A, Dhingra U, Kabole I, Deb S, Othman MK, Kabole FM. Effects of routine prophylactic supplementation with iron and folic acid on admission to hospital and mortality in preschool children in a high malaria transmission setting: community-based, randomised, placebo-controlled trial. Lancet. 2006 Jan 14;367(9505):133-43. doi: 10.1016/S0140-6736(06)67962-2. PMID 16413877
- [Background] Fawzi WW, Msamanga GI, Urassa W, Hertzmark E, Petraro P, Willett WC, Spiegelman D. Vitamins and perinatal outcomes among HIV-negative women in Tanzania. N Engl J Med. 2007 Apr 5;356(14):1423-31. doi: 10.1056/NEJMoa064868. PMID 17409323
- [Background] Tamura T, Yoshimura Y, Arakawa T. Human milk folate and folate status in lactating mothers and their infants. Am J Clin Nutr. 1980 Feb;33(2):193-7. doi: 10.1093/ajcn/33.2.193. PMID 7355792
- [Background] Khambalia A, Latulippe ME, Campos C, Merlos C, Villalpando S, Picciano MF, O'connor DL. Milk folate secretion is not impaired during iron deficiency in humans. J Nutr. 2006 Oct;136(10):2617-24. doi: 10.1093/jn/136.10.2617. PMID 16988136
- [Derived] Chowdhury R, Taneja S, Kvestad I, Hysing M, Bhandari N, Strand TA. Vitamin D status in early childhood is not associated with cognitive development and linear growth at 6-9 years of age in North Indian children: a cohort study. Nutr J. 2020 Feb 10;19(1):14. doi: 10.1186/s12937-020-00530-2. PMID 32041632
- [Derived] Kvestad I, Taneja S, Upadhyay RP, Hysing M, Bhandari N, Strand TA. Vitamin B12, Folate, and Cognition in 6- to 9-Year-Olds: A Randomized Controlled Trial. Pediatrics. 2020 Mar;145(3):e20192316. doi: 10.1542/peds.2019-2316. Epub 2020 Feb 4. PMID 32019814
- [Derived] Winje BA, Kvestad I, Krishnamachari S, Manji K, Taneja S, Bellinger DC, Bhandari N, Bisht S, Darling AM, Duggan CP, Fawzi W, Hysing M, Kumar T, Kurpad AV, Sudfeld CR, Svensen E, Thomas S, Strand TA. Does early vitamin B12 supplementation improve neurodevelopment and cognitive function in childhood and into school age: a study protocol for extended follow-ups from randomised controlled trials in India and Tanzania. BMJ Open. 2018 Feb 22;8(2):e018962. doi: 10.1136/bmjopen-2017-018962. PMID 29472265
- [Derived] Chowdhury R, Taneja S, Bhandari N, Kvestad I, Strand TA, Bhan MK. Vitamin-D status and neurodevelopment and growth in young north Indian children: a secondary data analysis. Nutr J. 2017 Sep 18;16(1):59. doi: 10.1186/s12937-017-0285-y. PMID 28923060
- [Derived] Kumar T, Taneja S, Sachdev HPS, Refsum H, Yajnik CS, Bhandari N, Strand TA; Study Group. Supplementation of vitamin B12 or folic acid on hemoglobin concentration in children 6-36 months of age: A randomized placebo controlled trial. Clin Nutr. 2017 Aug;36(4):986-991. doi: 10.1016/j.clnu.2016.07.002. Epub 2016 Jul 18. PMID 27486122
- [Derived] Kvestad I, Taneja S, Kumar T, Hysing M, Refsum H, Yajnik CS, Bhandari N, Strand TA; Folate and Vitamin B12 Study Group. Vitamin B12 and Folic Acid Improve Gross Motor and Problem-Solving Skills in Young North Indian Children: A Randomized Placebo-Controlled Trial. PLoS One. 2015 Jun 22;10(6):e0129915. doi: 10.1371/journal.pone.0129915. eCollection 2015. PMID 26098427
- [Derived] Strand TA, Taneja S, Kumar T, Manger MS, Refsum H, Yajnik CS, Bhandari N. Vitamin B-12, folic acid, and growth in 6- to 30-month-old children: a randomized controlled trial. Pediatrics. 2015 Apr;135(4):e918-26. doi: 10.1542/peds.2014-1848. PMID 25802345
- [Derived] Taneja S, Strand TA, Kumar T, Mahesh M, Mohan S, Manger MS, Refsum H, Yajnik CS, Bhandari N. Folic acid and vitamin B-12 supplementation and common infections in 6-30-mo-old children in India: a randomized placebo-controlled trial. Am J Clin Nutr. 2013 Sep;98(3):731-7. doi: 10.3945/ajcn.113.059592. Epub 2013 Jul 31. PMID 23902779